CLINICAL TRIAL: NCT05433246
Title: Effect of Massage Therapy on Peripheral Neuropathy and Life Quality of Colorectal Cancer wıth Patient Receiving Chemotherapy
Brief Title: Effects of Massage Therapy on Peripheral Neuropathy and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatma Arikan (Other)
Responsible Party: Sponsor-Investigator, Fatma Arikan, Assistant Professor, PhD, Akdeniz University
Organization: Akdeniz University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011/211
Record Dates: First submitted 2022-06-11; First posted 2022-06-27 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: Peripheral Neuropathy,; Chemotherapy; Massage; Life Quality; Colorectal Cancer
MeSH Terms: conditions — Peripheral Nervous System Diseases; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The patients received routine care.
- Massage therapy group (Experimental): The patients in the massage group were given classical massage for 2 consecutive days in each chemotherapy cycle (with an interval of two weeks). Massage therapy was performed with a classical massage technique using effleurage, petrissage, and superficial friction techniques for a total of 40 minutes on the areas below the elbow-forearm-hand (20 minutes), and below the knee-lower leg-foot (20 minutes). The patients in the massage group received 16 sessions of classical massage performed by the research nurse, who had classical massage training and certification.
  Interventions: Behavioral: Massage therapy group

INTERVENTIONS:
Behavioral: Massage therapy group — Massage therapy was performed with a classical massage technique using effleurage, petrissage, and superficial friction techniques for a total of 40 minutes on the areas below the elbow-forearm-hand (20 minutes), and below the knee-lower leg-foot (20 minutes). The patients in the massage group received 16 sessions of classical massage performed by the research nurse, who had classical massage training and certification.
  Arms: Massage therapy group

SUMMARY:
The aim of this randomized controlled experimental study was to determine the effect of massage applied to colorectal cancer patients receiving chemotherapy on peripheral neuropathy and quality of life.

DETAILED DESCRIPTION:
The aim of this randomized controlled experimental study was to determine the effect of massage applied to colorectal cancer patients receiving chemotherapy on peripheral neuropathy and quality of life.Investigation was carried out between February 2012- May 2013 with 52 patients meeting study criteria and receiving chemotherapy in Akdeniz University outpatient chemotherapy unit (28 study group, 24 control).

Massage therapy group:The experimental group patients were given a series of effleurage, petrissage and surface fraction types of classical massage on local parts of they're body-below, elbow-frontal arm-hand (20 minutes) and below knee-leg (lower part)-foot (20 minutes) two days of treatment of 16 times total.The patients in the massage group received 16 sessions of classical massage performed by the research nurse, who had classical massage training and certification.Baseline, patient characteristics , peripheral neuropathy symptoms, neuropathic pain, cancer and chemotherapy-related symptoms, and quality of life were completed. Peripheral neuropathy symptoms, cancer, and chemotherapy-related symptoms were assessed at each cycle (2th, 4th, 6th, 8th,10th,12th,14th, 16th. week- (two-week intervals)). Neuropathic pain and quality of life were measured at 4, 10, and 16 weeks. At week 16 (2 weeks after the intervention), the grade of peripheral sensory neuropathy was determined.

Control Group: The patients received routine care. Baseline, patient characteristics , peripheral neuropathy symptoms, neuropathic pain, cancer and chemotherapy-related symptoms, and quality of life were completed. Peripheral neuropathy symptoms, cancer, and chemotherapy-related symptoms were assessed at each cycle (2th, 4th, 6th, 8th,10th,12th,14th, 16th. week (two-week intervals)). Neuropathic pain and quality of life were measured at 4, 10, and 16 weeks. At week 16 (2 weeks after the intervention), the grade of peripheral sensory neuropathy was determined.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* have a diagnosis of colorectal cancer
* receiving FOLFOX-4 chemotherapy protocol
* to receive a maximum of 4 cycles of FOLFOX-4 chemotherapy
* platelet values over -100.000/mm3
* no obstacle to massage application

Exclusion Criteria:

* previously been diagnosed with polyneuropathy,
* has been diagnosed with diabetes,
* is addicted to alcohol,
* has been amputated at the extremities,
* has a skin infection and skin integrity disorder,
* has megaloblastic anemia, uses anticoagulants,
* takes drugs that hide or affect neuropathy findings
* has had massage therapy within the last month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2013-05-01 (Actual); Study Completion 2013-05-01 (Actual)

PRIMARY OUTCOMES:
Peripheral Neuropathy Evaluation Form | 16 week
  It was developed by the researcher by reviewing the literature in order to determine the symptoms of peripheral neuropathy in the upper and lower extremities of the patients (0=no symptoms, 4=very severe)
Self-Leeds Assessment of Neuropathic Symptoms and Signs Pain Scale (S-LANSS) | 16 weeks
  This scale measures neuropathic pain.The first five items of the scale show pain symptoms, while the last two items show allodynia and pinprick test self-report. A score of twelve points or more is considered as neuropathic pain (neuropathic pain yes:12 and higher).
MD Anderson Symptom Inventory | 16 weeks
  The scale includes symptoms (13 items), and measures how much the symptoms have interfered with six daily activities (general activity, mood, work, relations with others, walking, and enjoyment of life.) A high score indicates an increase in the severity of the symptom and negative impact on life. The rates the severity of symptoms with a score of 0-10, 0 "none" and 10 "as bad as you can imagine" over the past 24 hours.Interference is rated on a 0-10 numerical rating scale, 0 being "did not interfere" and 10 being "interfered completely." A score range of 5-6 is considered "moderate" and a range of 7-10 is considered "severe".
European Organisation for Research and Treatment of Cancer-Quality of Life Scale | 16 weeks
  It measures the quality of life of individuals diagnosed with cancer. This scale consists of three parts: general health, functional health and symptoms, and a total of 30 questions ((minimum score: 0 maximum score: 100).A high score indicates a high quality of life. Low scores on functional health (physical, role, emotional, cognitive, and social functions) and general health scales indicate poor quality of life. Low scores on the symptom subscale indicate higher quality of life.
American National Cancer Institute Cancer Therapy Evaluation Program Common Toxicity Criteria, Version 2.0 | 16 weeks
  It was used to grade Peripheral Neuropathy-sensory (minimum score: 0; maximum score: 4). Grade 0: Normal, no symptoms, Grade 4: permanent loss of sensation and impaired function. High grades indicate the height of the symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Feray Gökdogan, PhD, RN, Study Chair — Cyprus International University

IPD SHARING:
Plan to Share IPD: No